CLINICAL TRIAL: NCT01923909
Title: Comparison of Intraarticular Platelet-rich Plasma Injections With Intraarticular Corticosteroid Injections in the Treatment of Primary Knee Osteoarthritis : A Randomized Control Trial
Brief Title: Intraarticular Platelet-rich Plasma Injections Versus Corticosteroid Injections in Primary Knee Osteoarthritis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: King Hamad University Hospital, Bahrain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATF02092012
Record Dates: First submitted 2013-08-13; First posted 2013-08-16 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Osteoarthritis
Keywords: Knee; Osteoarthritis; Bahrain; PRP; Steroid; WOMAC; Oxford Knee Score; Platelet-rich plasma
MeSH Terms: conditions — Osteoarthritis | interventions — Pituitary Adenylate Cyclase-Activating Polypeptide; Methylprednisolone Acetate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intra-articular corticosteroid (Active Comparator): Intra-articular corticosteroid injections Patients receiving the IA corticosteroid will be injected 3mL of 0.5% Bupivacaine and 2mL of 80mg Depo Medrol in a 10cc syringe, using an aseptic technique into the suprapatellar pouch. After an IA corticosteroid injection, patients are always advised to rest for 24 hours, and weigh bear as little as possible for the following 3 days. The procedure will be performed by a senior resident with several years of experience or a consultant Orthopedic surgeon.
  Interventions: Drug: Intra-articular corticosteroid injections
- Intra-articular platelet-rich plasma (Experimental): IA PRP procedure This involves withdrawal of 10-15cc of patient's blood, which is collected and centrifuged in Rotofix 32 A Centrifuge machine at 1500 cycles/minute for 5 minutes. 3-4cc of the PRP is obtained and injected into the suprapatellar pouch using an aseptic technique. The procedure will be performed by the principal investigator, a qualified consultant Orthopedic surgeon. Analgesia will be administered as needed.
  Interventions: Drug: Intra-articular platelet-rich plasma

INTERVENTIONS:
Drug: Intra-articular platelet-rich plasma — Intra-articular platelet-rich plasma This involves withdrawal of 10-15cc of patient's blood, which is collected and centrifuged in Rotofix 32 A Centrifuge machine at 1500 cycles/minute for 5 minutes. 3-4cc of the PRP is obtained and injected into the supra patellar pouch using an aseptic technique. The procedure will be performed by the principal investigator, a qualified consultant Orthopedic surgeon. Analgesia will be administered as needed.
  Other Names: Prp
  Arms: Intra-articular platelet-rich plasma
Drug: Intra-articular corticosteroid injections — Patients receiving the IA corticosteroid will be injected 3mL of 0.5% Bupivacaine and 2mL of 80mg Depo Medrol in a 10cc syringe, using an aseptic technique into the supra patellar pouch. After an IA corticosteroid injection, patients are always advised to rest for 24 hours, and weigh bear as little as possible for the following 3 days. The procedure will be performed by a senior resident with several years of experience or a consultant Orthopedic surgeon.
  Other Names: Depo Medrol
  Arms: Intra-articular corticosteroid

SUMMARY:
Aim: To study and compare the clinical effects of platelet-rich plasma (PRP) injections and intra-articular (IA) corticosteroid injections in patients with primary osteoarthritis (OA) of the knee. This study aims to demonstrate this by using the Oxford Knee Score and Western Ontario and McMaster Universities Arthritis Index (WOMAC) to illustrate quantifiable difference between the two treatment modalities. Patient satisfaction will be compared by utilizing the Short-Form Survey-12 (SF-12) Score. Our null hypothesis states that intra-articular PRP injections is more beneficial in the long-term treatment of primary OA of the knee.

DETAILED DESCRIPTION:
This is a single blinded, randomized clinical trial. Subjects will be male or female patients with Grade 1,2 or 3 OA of the knee classified based on the radiological Kellgren -Lawrence grading system.

100 patients will be recruited for this study and 50 patients each will be randomized to one of the treatment groups using block randomization i.e. receiving either treatment IA corticosteroids or IA PRP injections. The patients will be informed of and will be consented to the treatment they will be receiving. An investigator from the research team, blinded to group assignment, will assist patients in completing the Oxford Knee score, WOMAC and SF-12 scores prior to receiving the treatment and at 6 weeks, 3 months and 6 months after receiving the treatment. In addition, they will be followed by regularly (at 3 weeks, 9 weeks, 4 months and 5 months) via telephone to inquire about any side effects of the treatment and to document patient satisfaction. Subjects in both groups will continue to receive concomitant treatments both pharmacological and nonpharmacological. All subjects will receive physiotherapy sessions with their respective intervention. Subjects will continue to receive treatment even if they wish to withdraw from the study at any point.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological diagnosis of Primary Osteoarthritis of Knee joint
* Grade 1, 2, or 3 as per Kellgren and Lawrence radiological grading system.
* Symptomatic at presentation as per Visual Analogue pain scale
* Above 18 years of age
* Consenting to participate

Exclusion Criteria:

* Deformities
* Malalignments
* Rheumatoid lesions
* Gouty lesions
* BMI more than 35
* Use of steroids in the recent 6 weeks
* Pregnant
* Breast feeding
* Active malignancy
* Active infections
* Hemoglobin less than 11
* Platelet less than 150,000/mm3 and
* Bleeding disorders/blood dyscrasias or hemoglobinopathies
* Any contraindications to treatments
* Uncontrolled diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in WOMAC Knee Score | 6 weeks to 6 months
  WOMAC - Western Ontario and Mcmaster index of Osteoarthritis

SECONDARY OUTCOMES:
Improvement in SF12 score | 6 weeks to 6 months
  SF12- patient satisfaction survey ( short form 12 point survey)
Improvement in Oxford Knee Score | 6 weeks to 6 months
  Oxford Knee Score

CONTACTS AND LOCATIONS:
Overall Officials: Ahsan J Butt, FRCS(T&O), Principal Investigator — King Hamad University Hospital; Tania Kumar, MBBCh, Principal Investigator — KHUH, RCSI-Bahrain; Fathima M Nasmy, MBBCh, Principal Investigator — KHUH, RCSI-Bahrain; Khaleefa ElMusharraf, MBBS,FRSPH, Principal Investigator — Royal College of Surgeons, Ireland; Fares Uddin, MBBCh, Principal Investigator — King Hamad University Hospital
Locations (1):
- Orthopedic Clinic King Hamad University Hospital, Al Muharraq, Bahrain